CLINICAL TRIAL: NCT01446861
Title: Pancreatic Failure in Patients With Cystic Fibrosis A Multimodal Study of Exocrine Pancreatic Failure in Cystic Fibrosis
Brief Title: Exocrine Pancreatic Function Testing in Cystic Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/2857-7
Record Dates: First submitted 2011-10-04; First posted 2011-10-05 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Pancreas; Exocrine function; Ultrasound; Contrast ultrasound
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Duodenal juice Serum, full Blood Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cystic fibrosis patients: Consecutive cystic fibrosis patients attending regular Controls at the CF clinic in Bergen
- Healthy controls: Age and gender matchet healthy Controls recruited by Board notice and advertising.

SUMMARY:
Purpose The purpose of this study is to develop and validate multimodal testing of exocrine pancreatic function (EPF). The investigators will be testing exocrine pancreatic function in patients with cystic fibrosis (CF). Exocrine pancreatic function and imaging will be correlated to age group, genotype, nutritional status and quality of life. Earlier detection of exocrine pancreatic failure in the non classical form of cystic fibrosis may be of therapeutically benefit.

Hypotheses Endoscopic short test can be applied in diagnosing and monitoring exocrine pancreatic function in patients with cystic fibrosis.

New functional testing of exocrine pancreatic function is superior to traditional testing with fecal elastase.

MRI and ultrasound methods can give volume output estimate in cystic fibrosis patients.

Contrast enhanced ultrasound can quantify reduced or delayed pancreatic perfusion and parenchymal changes in cystic fibrosis patients.

Elastography/ CEUS can be used in prediction and monitoring of fibrosis development and development of hepatocellular carcinoma in the liver of cystic fibrosis patients.

Immunohistochemical quantification of secretin/ cholecystokinin (CCK) producing cell in duodenum can be utilized as a model hormonal signaling in cystic fibrosis patients with exocrine pancreatic function.

DETAILED DESCRIPTION:
Study design: Observational, cohort studies.

Patient characterization: Age, gender, and Genetic status from electronical records.

Exocrine function testing (EPF): Secretin stimulated ultrasound and short endoscopic secretin test (EST). Faecal Elastase.

Imaging: Transabdominal ultrasound of the liver and pancreas. secretin stimulated MRI. Contrast enhanced ultrasound (CEUS) of the pancreas using SonoVue contrast.

Endpoints:

Study 1: Exocrine pancreatic function by duodenal bicarbonate/ Enzymes related to Genetics and F elastase.

Study 2: Ultrasound parenchymal changes of the pancreas related to Genetics and EPF.

Study 3/4: Pancreatic secretion by ultrasound, MRI and EST related to EPF Study 5; Perfusion of the pancreas by CEUS related to EPF

Study 6: Genotype-phenotype conciderations of the CF pancreas.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis cystic fibrosis. Age over 15 years. Assigned to routine control at department of lung diseases, Haukeland university hospital.

Exclusion Criteria:

* Unable to concent, allergies to Sonovue ultrasound contrast, pregnant or breastfeeding, contraindications against endoscopy.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cystic fibrosis patients over the age of 15 years Healthy controls between 18 and 67 years
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-01; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
peak lipase IE | one year

SECONDARY OUTCOMES:
enzyme production | 2 years

OTHER OUTCOMES:
emzyme production | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Georg Dimcevski, MD, PhD, Principal Investigator — Haukeland University Hospital; Odd H Gilja, Professor, Study Director — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Yes
Data will be published in peer rewieved journals